CLINICAL TRIAL: NCT00292513
Title: A Randomized Clinical Trial Comparing Tissue Adhesive (2-Octylcyanoacrylate) Vs. Absorbable Suture Vs. Non-Absorbable Suture for the Closure of Low Tension Facial and Neck Wounds in Children and Adolescents
Brief Title: Clinical Trial Comparing Tissue Adhesive Vs. Absorbable Suture Vs. Non-Absorbable Suture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rady Children's Hospital, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dermabond Study
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2005-05

CONDITIONS: Cyst of Face, Neck or Shoulder; Pilomatrixoma of Face, Neck or Shoulder

INTERVENTIONS:
Device: standard suture (5-0 prolene), topical skin adhesive (dermabond), absorbable suture (5-0 Chromic gut)

SUMMARY:
Standard suture is superior to both tissue adhesive (2-octyl cyanoacrylate) and absorbable sutures with respect to cosmetic outcome of, complication rate of and parental satisfaction with the closure of low tension facial, neck and shoulder, wounds in children and adolescents

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 18
* Pre-operative diagnosis of cyst or pilomatrixoma of neck, face or shoulder
* outpatient scheduled for outpatient or day surgery at Children's Hospital San Diego

Exclusion Criteria:

* known hypersensitivity to cyanoacrylate or formaldehyde
* lesions with any evidence of active infection or gangrene
* lesions on or across mucocutaneous surfaces
* lesions in which skin may be regularly exposed to body fluids
* lesions located in areas of dense natural hair (ie scalp)
* patients with peripheral vascular disease, insulin dependent diabetes mellitis or blood clotting disorders
* patients with known immunodeficiencies
* inability to return for follow-up

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bari B Cunningham, MD, Principal Investigator — Rady Children's Hospital, San Diego
Locations (1):
- Children's Hospital San Diego, San Diego, California, United States